CLINICAL TRIAL: NCT00611663
Title: VACCILUP "A Multicenter, Randomized Double-blind Trial Comparing Two Pneumococcal Vaccination Strategies in Patients With Systemic Lupus Erythematosus"
Brief Title: Safety Study of Two Vaccine Strategies in Patients With Systemic Lupus Erythematosus
Acronym: VACCILUP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060241
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Pneumococcal vaccine; SLE; Vaccination; Immunosuppression; SLE as defined by the ACR classification; Stable SLE; SLE treated by systemic corticosteroids
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vaccination with conjugate vaccine Prevenar® (WYETH-LEDERLE) at week 0 and Poly Saccharidic vaccine Pneumo23® (Sanofi Pasteur MSD) after 6 months (W24)
  Interventions: Biological: Prevenar® and Pneumo23®
- 2 (Placebo Comparator): Vaccination with placebo at W0 and Poly Saccharidic vaccine Pneumo23® at W24
  Interventions: Biological: Placebo, Pneumo23®

INTERVENTIONS:
Biological: Prevenar® and Pneumo23® — Vaccination with conjugate vaccine Prevenar® (WYETH-LEDERLE)at week 0 and Poly Saccharidic vaccine Pneumo23® (Sanofi Pasteur MSD) after 6 months (W24)versus2)
  Arms: 1
Biological: Placebo, Pneumo23® — Vaccination with placebo at W0 and Poly Saccharidic vaccine Pneumo23® at W24
  Arms: 2

SUMMARY:
The aim of this study is to compare the immunological efficacy of two pneumococcal vaccination strategies in patients with systemic lupus erythematosus (SLE) treated with corticosteroids associated or not with other immunosuppressive drugs : 1) a prime-boost strategy using vaccination with conjugate vaccine (Prevenar®) at week 0 and Poly Saccharidic vaccine (Pneumo23®) after 6 months (W24)2) compared to the standard vaccination with Poly Saccharidic vaccine (Pneumo23®) at W24 after placebo at W0

DETAILED DESCRIPTION:
Infections are more frequent and potentially more serious in patients with SLE compared to healthy subjects. This risk increases when patients are treated with corticosteroids and/or immunosuppressive drugs.Among serious infections which can happen in this context, respiratory infections are among the most frequent and Streptococcus pneumoniae is one of the most often responsible germs.Although there are no specific study in SLE, these findings indicate that patients with SLE could benefit from a preventive vaccination against pneumococcal infections.Two pneumococcal vaccines are available: Pneumo23®, a Poly Saccharidic vaccine indicated for adults and children > 2 years at risk of pneumococcal infections; and Prevenar®, a conjugate vaccine, indicated for children < 2 years.Pneumo23® has been found to be safe in SLE but less immunogenic than in general population.Prevenar® has already been studied in immunocompromised patients (HIV-infected patients, patients after renal transplantation). It has been shown that immunological efficacy is better when Prevenar® is administrated prior to Pneumo23®, compared to Pneumo23® administrated alone.To our knowledge, this prime-boost strategy has not been assessed in patients with SLEThe primary objective of the study is to compare immunological efficacy of two pneumococcal vaccination strategies in patients with systemic lupus erythematosus (SLE) treated with corticosteroids associated or not with other immunosuppressive drugs : 1) Vaccination with conjugate vaccine (Prevenar®) at week 0 and Poly Saccharidic vaccine (Pneumo23®) after 6 months (W24)2) Vaccination with placebo at W0 and Poly Saccharidic vaccine (Pneumo23®) at W24Secondary objectives are:

* To compare the clinical and biological tolerance of the two vaccinal strategies·
* To evaluate the durability of sero protection at 6 and 24 months after vaccination by Pneumo23®
* To search predictive factors determinant of the pneumococcal vaccine response

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* SLE as defined by the ACR classification
* Stable SLE (treatment not modified during the 2 months preceding the inclusion date W0)
* SLE treated by immunosuppressant only or systemic corticosteroids at a dose ≥ 5 mg/j or systemic corticosteroids at any dose associated with one or more immunosuppressive drugs
* SLE treated by hydroxychloroquine only
* 31 months following
* females must have an effective method of contraception during the first 7 months of the study and with a negative serum or urinary pregnancy test
* females not wishing to have a child during the 7 months following W0
* physical examination
* signed written and informed consent

Exclusion Criteria:

* pregnant females or females wishing to have a child during the 7 months following W0
* subjects infected with HIV and/or HBV( Ag HBs+) and or HVC
* medical history of allergy to any vaccine component
* receipt of any pneumococcal vaccine less than 5 years
* receipt of other vaccine within one month prior to enrolment (inclusion visit W0)
* receipt of immunoglobulin within three months prior to enrolment (inclusion visit W0)
* splenectomy
* hematopoietic disorders which give contra-indications to intramuscular and hypodermic route injections,
* active malignancy , cirrhosis
* intercurrent illness within one month prior to enrolment (inclusion visit W0)
* patients under biotherapy (anti-CD20)must not been included if the interval between vaccination and the end of the biotherapy is less than one year.
* participation to another clinical study during the first 7 months of the study
* subject not covered by Health Insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-05; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of responders for more than 5 serotypes among the 7 serotypes common between conjugate and Poly Saccharidic vaccines (ie. serotypes 4, 6B, 9V, 14, 18C, 19F and 23F). | 31 months

SECONDARY OUTCOMES:
Proportion of patients presenting a disease exacerbation(defined as an increase of ³3 points on the SLEDAI score and/or need to increase treatment with corticosteroids or immunosuppressive drugs) during the 12 months following the first vaccination | 13 months
Proportion of patients with local or systemic reactions following vaccination | 31 months
Comparison of serum antibodies titers obtained at W28 for each of the tested serotypes | 28 weeks
Comparison of ELISA persistent responses six months and 2 years after vaccination with Pneumo23® (M12 and M30) | 12 months + 30 months
Research of predictive factors of immunological response disease activity at M0 (defined by SLEDAI), SLE treatment and others variables witch can affect the response. | 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, PhD, Principal Investigator — CIC vaccinologie Cochin Hospital
Locations (1):
- CIC Vaccinologie - Hopital Cochin, Paris, France

REFERENCES:
- [Background] Grabar S, Groh M, Bahuaud M, Le Guern V, Costedoat-Chalumeau N, Mathian A, Hanslik T, Guillevin L, Batteux F, Launay O; VACCILUP study group. Pneumococcal vaccination in patients with systemic lupus erythematosus: A multicenter placebo-controlled randomized double-blind study. Vaccine. 2017 Sep 5;35(37):4877-4885. doi: 10.1016/j.vaccine.2017.07.094. Epub 2017 Aug 4. PMID 28784280